CLINICAL TRIAL: NCT03703934
Title: Central Pain Mechanisms in Patients With Hand-Osteoarthritis, Psoriatic Arthritis and Healthy Controls
Status: Suspended | Type: Observational
Why Stopped: COVID-19
Sponsor: Aalborg University Hospital (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Principal Investigator, Jonathan Vela, Medical Doctor, Aalborg University Hospital
Other Study IDs: 210417
Record Dates: First submitted 2018-10-01; First posted 2018-10-12 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Arthritis, Psoriatic; Hand Osteoarthritis
Keywords: Pain phenotyping; Quantitative sensory testing
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Psoriatic Arthritis: Patients with painful psoriatic arthritis
- Hand Osteoarthritis: Patients with painful nodal non-erosive hand osteoarthritis
- Healthy Controls: Patients without a painful condition

SUMMARY:
In this trial different parts of the pain signalling system involved in two rheumatic diseases - painful hand osteoarthritis and psoriatic arthritis, is examined. These measurements will be compared to those of healthy volunteers

The hypothesis is that patients with hand osteoarthritis and psoriatic arthritis react differently to painful and non-painful stimuli compared with the healthy volunteers.

The aim is to recruit 66 patients with painful hand-osteoarthritis, 66 patients with painful psoriatic arthritis and 66 healthy subjects not currently suffering from any pain conditions.

After completing an informed consent form subjects will participate in a single clinical visit. The pain signalling system is examined using pressure algometry and cuff algometry. A pressure algometer is a pistol shaped device that elicits pressure through a rod and a cuff algometer is akin to a blood pressure cuff. Different thresholds will be measured, such as when the sensation of pressure becomes painful and when the painful pressure becomes unbearable.

Participants will also get hand strength tested, have their joints examined and answer questionnaires regarding daily function and quality of life.

Furthermore participants will get blood drawn which is analysed for the presence of markers of inflammation and joint degeneration.

DETAILED DESCRIPTION:
Purpose and rationale for this study:

Treating painful hand osteoarthritis (Hand-OA) and psoriatic arthritis (PsA) is a clinical challenge because the exact pain mechanisms remain unknown. Both conditions seem to involve both central and peripheral pain mechanisms and inflammation to some degree. However, it remains unknown whether the pain mechanisms are homogenous among patients with said conditions or if different pain phenotypes exist that may respond differently to treatments.

The initiative on Methods, Measurement, and Pain Assessment in Clinical Trials (IMMPACT) consortium has recognized this. IMMPACT recommends that clinical trials with chronic pain patients assess different domains of the pain experience (psychosocial, pain qualities, sleep, and pain pathways) to examine if pain phenotypes exist and whether different treatment modalities are more effective for certain phenotypes.

Methods: A cross-sectional study examining the difference in pain phenotype and pain mechanisms between patients with Hand-OA, PsA and healthy pain free controls using questionnaire assessments and quantitative sensory testing aiming at investigating pain pathways in the central nervous system. Participants will also have blood drawn to evaluate serological biomarkers for inflammation and joint degeneration.

Aim: To examine the pain phenotypes and assess differences in pressure pain threshold between patients with Hand-OA, PsA and healthy pain free controls.

Patients and controls: Patients with nodal non-erosive Hand-OA or PsA and visual analogue scale for pain (VAS pain) during the last 24hours of 30mm or more.

Controls are healthy age and gender matched subjects with no known chronic pain conditions and maximal pain during last 24 hours under 10mm on a 100mm VAS.

Examination programme: All participants will receive a full medical interview and a physical examination which includes auscultation, blood pressure, heart rate and saturation measurements and BMI calculation. All participants will have blood drawn for later examination for markers of inflammation and degeneration. All participants will go through Quantitative Sensory Testing (QST). QST covers a wide range of different examinations techniques used to assess the functional status of the somatosensory system33. In the present study pressure algometry and cuff algometry will be performed.

Pain phenotyping: Participants will answer a series of questionnaires related to the pain experience to assess: Anxiety and depression (the hospital anxiety and depression scale), pain catastrophizing (the pain catastrophizing scale), pain description (The short form McGill questionnaire and pain detect questionnaire), sleep quality (Pittsburgh sleep quality index) and a widespread pain assessment questionnaire. To assess function and quality of life the Short form 36 and Health assessment questionnaire will be used.

Patients with PsA: Will receive an examination for disease specific tests including: joint tenderness and swelling using the European league against rheumatism (EULAR) 66/68 regiment, dactylitis evaluation using Leeds dactylitis index basic, skin involvement using the psoriasis area and severity index and nail psoriasis via nail psoriasis severity index.

Patients with Hand-OA: Will receive the following disease specific examinations evaluation of tender and swollen joints of the hands and wrists. Grip and pinch strength measurements using a hand-held dynamometer.

ELIGIBILITY:
Inclusion criteria Hand-OA

* Patients (above 18 years) with Hand-OA according to the American Collage of Rheumatology (ACR) criteria (1990)
* Hand-OA of the phenotype: Nodal, Non-erosive.
* Ability and willingness to give written informed consent and to meet the requirements of the study protocol.
* VAS pain during the last 24 hours 30mm or more
* Negative pregnancy test (serum HCG) prior to trial start (for women of childbearing potential) and the use of contraception throughout the study period and for 3 months after conclusion of the study period for males and females of childbearing potential. The forms of contraception include: intrauterine device (IUD) and hormonal contraceptives (contraceptive pill, implant, patch or injection or vaginal ring). Sterile and non-fertile participants do not have to use contraception. Sterile or non-fertile is defined as having undergone surgical sterilization (vasectomy / bilateral tubectomy, hysterectomy or bilateral oophorectomy) or post-menopausal status, defined as absence of menstrual period for at least 12 months prior to enrollment.

Inclusion criteria PsA

* Patients (over 18 years) with PsA according to the Clarification Criteria for Psoriatic Arthritis (CASPAR) criteria (2006)
* Ability and willingness to give written informed consent and to meet the requirements of the study protocol.
* VAS pain during the last 24 hours 30mm or more
* Negative pregnancy test (serum human chorionic gonadotropin (HCG)) prior to trial start and the use of contraception throughout the study period and for 1 month after conclusion of the study period for women of childbearing potential. The forms of contraception include: intrauterine device (IUD) and hormonal contraceptives (contraceptive pill, implant, patch or injection or vaginal ring). Sterile and non-fertile participants do not have to use contraception. Sterile or non-fertile is defined as having undergone surgical sterilization (vasectomy / bilateral tubectomy, hysterectomy or bilateral oophorectomy) or post-menopausal status, defined as absence of menstrual period for at least 12 months prior to enrollment.

Inclusion criteria healthy controls

* Men and women age over18 years
* Ability and willingness to give written informed consent and to meet the requirements of the study protocol.

Exclusion Criteria:

* Other known inflammatory rheumatic disease (i.e. rheumatoid arthritis, gout) *
* Erosive Hand-OA (One or more erosive joints on plain x-ray)
* Isolated Hand-OA of the first metacarpal joint or this joint as the most painful*
* Other known pain condition (i.e. fibromyalgia, Carpel tunnel syndrome, polyneuropathy)
* Other known disease where exacerbations need to be treated with systemic corticosteroids (i.e. certain types of inflammatory bowl disease) or patients who have received systemic corticosteroid treatment during the last 3 months.
* Planning pregnancy, pregnant or breastfeeding. (Fertile women will be tested for pregnancy)
* Planned major surgery or recent major surgery (last 8weeks)
* Verified malignant disease
* History of epilepsy or severe cramps
* History of serious cardiovascular pathology
* Lacking ability to corporate with the research staff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: PsA and Hand-OA patients will be picked from primary and secondary care. Healthy volunteers will be picked from the community.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2018-10-20 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Between group difference in Pressure pain threshold (PPT) | Day One
  Difference PPT between groups measured in kPa

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rheumatology Aalborg Universityhospital North, Aalborg, Denmark